CLINICAL TRIAL: NCT00610428
Title: A Multi-center, Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of StaccatoTM Prochlorperazine for Inhalation in Patients With Migraine Headache
Brief Title: Staccato Prochlorperazine in Migraine (in Clinic)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-001-201
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2008-01

CONDITIONS: Migraine Headache, With or Without Aura
Keywords: Migraine, Staccato Prochlorperazine; Migraine headache with or without aura.
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inhaled Placebo (Placebo Comparator): Inhaled Staccato Placebo
  Interventions: Drug: Staccato Placebo
- Inhaled PCZ 5 mg (Experimental): Inhaled Staccato Prochlorperazine 5 mg
  Interventions: Drug: Staccato Prochlorperazine 5 mg
- Inhaled PCZ 10 mg (Placebo Comparator): Inhaled Staccato Prochlorperazine 10 mg
  Interventions: Drug: Staccato Prochlorperazine 10 mg

INTERVENTIONS:
Drug: Staccato Placebo — Inhaled Staccato Placebo
  Arms: Inhaled Placebo
Drug: Staccato Prochlorperazine 5 mg — Inhaled Prochlorperazine 5 mg
  Arms: Inhaled PCZ 5 mg
Drug: Staccato Prochlorperazine 10 mg — Inhaled Prochlorperazine10 mg
  Arms: Inhaled PCZ 10 mg

SUMMARY:
Development of Staccato Prochlorperazine for the treatment of migraine headache.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have migraine headache with or without aura (diagnosis according to International Headache Society guidelines) for at least 6 months, who have been pain free for at least 48 hours since the end of their last migraine attack, who have a pain rating of Moderate or Severe prior to dosing.

Exclusion Criteria:

* Subjects who have taken any other migraine or pain medication within 48 hours of randomization, with a history of allergy or intolerance to phenothiazines and related drugs, or are considered by the investigator, for any reason, to be an unsuitable candidate for receiving prochlorperazine, or unable to use the inhalation device, must be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheena Auroa, MD, Principal Investigator; Roger K Cady, MD, Principal Investigator; Arthur Elkind, MD, Principal Investigator; Fred Freitag, DO, Principal Investigator; Lisa Mannix, MD, Principal Investigator; Niana T Mathew, MD, Principal Investigator; Egilius LH Spierings, MD, Principal Investigator; Stewart Tepper, MD, Principal Investigator
Locations (1):
- Arthur H. Elkind, MD, Mount Vernon, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Background] Avram MJ, Spyker DA, Henthorn TK, Cassella JV. The pharmacokinetics and bioavailability of prochlorperazine delivered as a thermally generated aerosol in a single breath to volunteers. Clin Pharmacol Ther. 2009 Jan;85(1):71-7. doi: 10.1038/clpt.2008.184. Epub 2008 Oct 1. PMID 18830225

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inhaled Placebo | Inhaled PCZ 5 mg | Inhaled PCZ 10 mg
Started | 24 | 24 | 27
Completed | 24 | 23 | 25
Not Completed | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Placebo | Inhaled PCZ 5 mg | Inhaled PCZ 10 mg | Total
Number analyzed (Participants) | 24 | 24 | 27 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 27 | 75
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11.4) | 43.6 (10.8) | 41.9 (10.1) | 43.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 23 | 58
  Male | 9 | 4 | 4 | 17
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 27 | 75

OUTCOME MEASURES:

1. Primary Outcome: Headache Pain Relief at 2 hr Post-dose by 2-point Definition
Description: patient headache pain relief defined as a 2 point reduction as measured on the scale: 0=NO headache pain, 1 = MILD headache pain, 2 = MODERATE headache pain, 3 = SEVERE headache pain
Time Frame: 2 hours after treatment
Population: ITT Population with LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo | Inhaled PCZ 5 mg | Inhaled PCZ 10 mg
Number analyzed (Participants) | 24 | 24 | 27
Participants | 6 | 11 | 13

2. Secondary Outcome: Survival Analysis for Time to Pain Relief
Description: Survival Analysis for Time to the First Success Based on Pain Relief by 2-Point Definition
Time Frame: from treatment (time = 0) to 2 hours post treatment
Population: ITT Population by Treatment Assigned
Measure: Mean (Standard Error); unit: minutes to pain relief
Arm/Group | Inhaled Placebo | Inhaled PCZ 5 mg | Inhaled PCZ 10 mg
Number analyzed (Participants) | 24 | 24 | 27
minutes to pain relief | 115.4 (4.92) | 96.5 (8.22) | 88.6 (8.33)
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled PCZ 5 mg; Survival time is defined as time to the first successful headache relief; Test type: Superiority; p = 0.0840, Survival — p-values calculated by Log-rank Test in step-down sequence (10 mg to 5 mg)
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled PCZ 10 mg; Test type: Superiority — Survival time is defined as time to the first successful headache relief; p = 0.0383, Survival — p-values calculated by Log-rank Test in step-down sequence (10 mg to 5 mg)

ADVERSE EVENTS:
Time Frame: From informed consent through 30 days after last treatment
Description: Adverse events (AE) observed by the Investigator or study personnel during study assessments and throughout post-dosing period or when volunteered by the patient regardless of treatment group or suspected causal relationship to study drugs were recorded on the AE CRF. The severity of the AE and relationship to study drug was determined by the investigator.
Arm/Group | Inhaled Placebo | Inhaled PCZ 5 mg | Inhaled PCZ 10 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 8/24 | 12/24 | 16/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo (N=24) | Inhaled PCZ 5 mg (N=24) | Inhaled PCZ 10 mg (N=27)
Lacrimation Increased (Eye disorders) | 2 (2) | 1 (1) | 3 (3)
Dysgeusia (Gastrointestinal disorders) | 2 (2) | 7 (7) | 5 (5)
Somnolence (Nervous system disorders) | 2 (2) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 2 (2)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less